CLINICAL TRIAL: NCT05291637
Title: Endovascular Therapy vs Medical Management of PosterIor Cerebral Artery Occlusion Stroke
Brief Title: Posterior cerebraL ArTery Occlusion Study
Acronym: PLATO
Status: Completed | Type: Observational
Sponsor: Boston Medical Center (Other)
Collaborators: Heidelberg University (Other)
Responsible Party: Sponsor
Other Study IDs: H-40712
Record Dates: First submitted 2022-03-04; First posted 2022-03-22 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Stroke, Acute Ischemic
Keywords: Posterior occlusion artery (PCA); Intravenous thrombolysis (IVT); Endovascular therapy (EVT); Modified Rankin Scale (mRS)
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Medical management cohort: Patients who have undergone medical management stroke treatment from 1/01/2003 to 01/01/2022; this could include intravenous thrombolysis.
- EVT management cohort: Patients who have undergone EVT stroke treatment from 01/01/2015 to 01/01/2022

SUMMARY:
For this retrospective study, the investigators will collect and analyze data of patients who presented with posterior artery occlusion and underwent mechanical thrombectomy (the type of endovascular stroke treatment) and intravenous thrombolysis (the type of non-endovascular stroke treatment).

The electronic health records will be queried for the demographic, medical history, and outcomes data of all patients with posterior cerebral artery occlusion who underwent mechanical thrombectomy, intravenous thrombolysis (IVT), or medical management.

DETAILED DESCRIPTION:
The primary aims of the research are to evaluate, in patients presenting with posterior artery occlusion (PCA), whether favorable outcome would be superior for EVT compared to Medically Management (MM), inclusive of intravenous thrombolysis (IVT), as measured by:

* 90-day modified Rankin Scale (mRS) ordinal shift or
* decrease in NIH Stroke Scale/Score (NIHSS) by two points at 24 hours or at hospital discharge

The secondary aims are to evaluate in patients presenting with PCA occlusion, other outcome and safety metrics:

* 90-day functional independence, mRS 0-2
* 90-day excellent outcome, mRS 0-1
* Visual field recovery (none, partial, complete) by 90-days
* rate of reperfusion by modified thrombolysis in cerebral infarction (TICI) scale grade
* any intracranial hemorrhage
* symptomatic intracranial hemorrhage
* mortality

In subgroup analysis, the investigators aim to identify subgroups that may confer differential treatment benefit by:

* location of occlusion on the PCA segment (P1, P2, P3)
* NIHSS strata (0-6, 7-15,>16)
* time from symptom onset to treatment (0 to <6h vs 6-24h)
* posterior circulation (PC) Acute Stroke Prognosis Early Computed Tomography Score (ASPECTS)
* visual field defect on presentation

The investigators hypothesize that greater benefit in outcomes would be seen in EVT treated patients with higher NIHSS, more proximal PCA occlusion, higher PC ASPECTS scores, and shorter time from symptom onset to treatment.

ELIGIBILITY:
Inclusion Criteria:

* Had an ischemic stroke with isolated posterior cerebral artery occlusion (P1, P2, or P3 segments) and was medically managed or managed with EVT during the study time period.

Exclusion Criteria:

* Patient with documented basilar artery occlusion and concomitant PCA occlusion
* Patient with documented basilar artery occlusion, migration with secondary PCA occlusion

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients identified from electronic health records who have undergone stroke medical management treatment from 1/01/2003 to 01/01/2022 and patients who have undergone EVT stroke treatment from 01/01/2015 - 01/01/2022.
Sampling Method: Non-Probability Sample
Enrollment: 1282 (Actual)
Dates: Start 2022-01-05 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Change in stroke outcome based on modified Rankin Scale (mRS) | baseline, 90 days
  The Modified Rankin Scale (mRS) assesses disability in patients who have suffered a stroke and is compared over time to check for recovery and degree of continued disability. Scores can range from 0-6, where 0 is no disability, 5 is disability requiring constant care for all needs, and 6 is death. For this outcome an ordinal shift analysis will be done, assessing all changes across the range from baseline at 90 days.
Change in NIH Stroke Score (NIHSS) | baseline, 7 days
  The NIH Stroke Scale/Score (NIHSS) is is a 15-item neurologic examination stroke scale used to evaluate the effect of acute cerebral infarction on the levels of consciousness, language, neglect, visual-field loss, extraocular movement, motor strength, ataxia, dysarthria, and sensory loss. Scores can range from 0 to 42 and higher scores are associated with more severe stroke: 1-4= Minor stroke, 5-15= Moderate stroke, 15-20= Moderate/severe stroke, and 21-42 =Severe stroke.

CONTACTS AND LOCATIONS:
Overall Officials: Thanh N Nguyen, MD, Principal Investigator — Boston Medical Center, Neurology; Simon Nagel, MD, Principal Investigator — Heidelberg University Hospital, Neurology
Locations (22):
- United States (9):
  - University of Miami, Miami, Florida
  - Miami Baptist Health, Miami, Florida
  - Emory University School of Medicine, Atlanta, Georgia
  - Boston Medical Center, Boston, Massachusetts
  - Cooper University Healthcare, Camden, New Jersey
  - University of Buffalo, Buffalo, New York
  - Mount Sinai Health, New York, New York
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - UT Texas Medical Center, Houston, Texas
- Helsinki University Hospital, Helsinki, Finland
- Germany (6):
  - Charite Berlin, Berlin
  - Universitätsklinikum Knappschaftskrankenhaus Bochum, Bochum
  - University Clinics Dresden, Dresden
  - Universitätsklinikum Erlangen, Erlangen
  - University Medical Center Hamburg-Eppendorf, Hamburg
  - Heidelberg University, Heidelberg
- IRCCS Istituto delle Scienze Neurologiche di Bologna, Bologna, Italy
- Portugal (2):
  - Egas Moniz Hospital, Lisbon
  - Centro Hospitalar Universitário de Lisboa Central, Lisbon
- Vall D'Hebron, Barcelona, Spain
- Switzerland (2):
  - Lausanne University Hospital, Lausanne, Canton of Vaud
  - University Hospital Basel, Basel

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Herweh C, Abdalkader M, Nguyen TN, Puetz V, Schone D, Kaiser D, Chen CH, Jeng JS, Mohlenbruch MA, Ringleb PA, Nagel S. Mechanical Thrombectomy in Isolated Occlusion of the Proximal Posterior Cerebral Artery. Front Neurol. 2021 Jul 29;12:697348. doi: 10.3389/fneur.2021.697348. eCollection 2021. PMID 34393977
- [Background] Berberich A, Finitsis S, Strambo D, Michel P, Herweh C, Meyer L, Hanning U, Strbian D, Abdalkader M, Nogueira RG, Puetz V, Kaiser DPO, Olive-Gadea M, Ribo M, Fragata I, Marto JP, Romoli M, Ringleb PA, Nguyen TN, Nagel S. Endovascular therapy versus no endovascular therapy in patients receiving best medical management for acute isolated occlusion of the posterior cerebral artery: A systematic review and meta-analysis. Eur J Neurol. 2022 Sep;29(9):2664-2673. doi: 10.1111/ene.15410. Epub 2022 Jun 17. PMID 35587104
- [Result] Nguyen TN, Qureshi MM, Strambo D, Strbian D, Raty S, Herweh C, Abdalkader M, Olive-Gadea M, Ribo M, Psychogios M, Fischer U, Nguyen A, Kuramatsu JB, Haupenthal D, Kohrmann M, Deuschl C, Kuhne Escola J, Yaghi S, Shu L, Puetz V, Kaiser DPO, Kaesmacher J, Mujanovic A, Marterstock DC, Engelhorn T, Klein P, Haussen DC, Mohammaden MH, Abdelhamid H, Souza Viana L, Cunha B, Fragata I, Romoli M, Diana F, Virtanen P, Lappalainen K, Clark J, Matsoukas S, Fifi JT, Sheth SA, Salazar-Marioni S, Marto JP, Ramos JN, Miszczuk M, Riegler C, Jadhav AP, Desai SM, Maus V, Kaeder M, Siddiqui AH, Monteiro A, Masoud HE, Suryadevara N, Mokin M, Thanki S, Siegler JE, Khalife J, Linfante I, Dabus G, Asdaghi N, Saini V, Nolte CH, Siebert E, Meinel TR, Finitsis S, Mohlenbruch MA, Ringleb PA, Berberich A, Nogueira RG, Hanning U, Meyer L, Michel P, Nagel S. Endovascular Versus Medical Management of Posterior Cerebral Artery Occlusion Stroke: The PLATO Study. Stroke. 2023 Jul;54(7):1708-1717. doi: 10.1161/STROKEAHA.123.042674. Epub 2023 May 24. PMID 37222709
- [Result] Strambo D, Michel P, Nguyen TN, Abdalkader M, Qureshi MM, Strbian D, Herweh C, Mohlenbruch MA, Raty S, Olive-Gadea M, Ribo M, Psychogios M, Fischer U, Nguyen A, Kuramatsu JB, Haupenthal D, Kohrmann M, Deuschl C, Kuhne Escola J, Demeestere J, Lemmens R, Vandewalle L, Yaghi S, Shu L, Puetz V, Kaiser DPO, Kaesmacher J, Mujanovic A, Marterstock DC, Engelhorn T, Requena M, Dasenbrock HH, Klein P, Haussen DC, Mohammaden MH, Abdelhamid H, Souza Viana L, Cunha B, Fragata I, Romoli M, Diana F, Hu W, Zhang C, Virtanen P, Lauha R, Jesser J, Clark J, Matsoukas S, Fifi JT, Sheth SA, Salazar-Marioni S, Marto JP, Ramos JN, Miszczuk M, Riegler C, Poli S, Poli K, Jadhav AP, Desai SM, Maus V, Kaeder M, Siddiqui AH, Monteiro A, Masoud HE, Suryadareva N, Mokin M, Thanki S, Alpay K, Ylikotila P, Siegler JE, Linfante I, Dabus G, Asdaghi N, Saini V, Nolte CH, Siebert E, Serrallach BL, Weyland CS, Hanning U, Meyer L, Berberich A, Ringleb PA, Nogueira RG, Nagel S. Endovascular Versus Medical Therapy in Posterior Cerebral Artery Stroke: Role of Baseline NIHSS Score and Occlusion Site. Stroke. 2024 Jul;55(7):1787-1797. doi: 10.1161/STROKEAHA.124.047383. Epub 2024 May 16. PMID 38753954
- See also: Endovascular Thrombectomy Versus Intravenous Thrombolysis of Posterior Cerebral Artery Occlusion Stroke — https://j-stroke.org/journal/view.php?number=533